CLINICAL TRIAL: NCT04513938
Title: Interest of the Second Phase of the Oral Challenge Test in Patients With Suspected Long-standing Penicillin Allergy
Acronym: PENI
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PENI
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Allergy Penicillin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The most common drug allergy reported is penicillin allergy, approximately 10% of the world's population. According to the latest studies, only 1-2% of them have a proven hypersensitivity to penicillins. Being wrongly labeled "allergic" leads to a loss of chance for patients to be treated with a molecule of less efficacy than penicillins, an increase in bacterial resistance by broadening the spectrum of action of the molecules prescribed as an alternative and ultimately a additional financial cost. There are several forms of hypersensitivity: the two most classic: immediate hypersensitivity (type I according to Gell and Combs) with a reaction within an hour of taking and non-immediate hypersensitivity with a reaction occurring several days later (type IV according to Gell and Combs). A large majority of patients report a history of allergy in childhood that is poorly described and most often absent from health records. In most cases, this may be a viral rash concomitant with a febrile episode mistakenly mistaken for an allergic skin reaction. Patients are then tested for several decades, in adulthood, after their initial reaction. This latency of time involves a risk of negativation of the allergic tests and it is not excluded that the skin tests or drug reintroductions re cause sensitization to the antibiotic tested and that ultimately the patient reacts when taking the future drug. In fact, it is recommended to optimally explore patients approximately 6 months after an allergic reaction (except for severe drug eruptions).

The exploration of drug hypersensitivity to penicillins therefore involves a strict questioning of the circumstances of the so-called allergic reaction allowing the reaction to be classified as immediate or delayed, then skin tests (prick test, IDR and Patch test according to the immediate profile or delayed) and finally the hospital provocation test. While provocation tests are carried out conventionally most often within one day, it has been shown that some patients react several days after taking penicillin repeatedly: 6.1% have a reaction in their protocol of taking for 5 days at home in the context of a delayed allergy.

In the allergology service at hôpital Paris Saint-Joseph, the protocol corresponds to 2 successive reintroductions.

This study is to evaluate the protocol for reintroducing Amoxicillin or Augmentin carried out over two stages: a first with 100 mg (i.e. 1 / 10th of a dose) then a second with a dose of 1200 mg 1 month later. It would be a question of seeing if with the second reintroduction, one could not catch up with allergic people who would have presented a false negative during the first reintroduction because of explorations too far away from their initial reaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patient with a history of drug allergy and eviction for more than 12 months of penicillins A: mainly amoxicillin and amoxicillin + clavulanic acid
* Patients who had two amoxicillin or Augmentin Oral Challenge Test between December 2017 and December 2018 in allergology department of the Paris Saint-Joseph hospital
* French-speaking patient

Exclusion Criteria:

* Patient with uncontrolled asthma
* Patient with an ongoing infection
* Patient with positive skin tests for penicillin before the first TPO
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient objecting to participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be carried out on the data of patients, having carried out two TPO of amoxicillin or Augmentin between December 2017 and December 2018 in HDJ or during an allergology consultation within the Paris Saint-Joseph hospital.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the second oral challenge test | Day 1
  This outcome corresponds to the percentage of patients diagnosed with allergies during the second Oral Challenge Test versus all patients with a negative first Oral Challenge Test.

CONTACTS AND LOCATIONS:
Overall Officials: GEST Noemie, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Solensky R, Earl HS, Gruchalla RS. Lack of penicillin resensitization in patients with a history of penicillin allergy after receiving repeated penicillin courses. Arch Intern Med. 2002 Apr 8;162(7):822-6. doi: 10.1001/archinte.162.7.822. PMID 11926858
- [Result] Marwood J, Aguirrebarrena G, Kerr S, Welch SA, Rimmer J. De-labelling self-reported penicillin allergy within the emergency department through the use of skin tests and oral drug provocation testing. Emerg Med Australas. 2017 Oct;29(5):509-515. doi: 10.1111/1742-6723.12774. Epub 2017 Apr 5. PMID 28378949
- [Result] Shenoy ES, Macy E, Rowe T, Blumenthal KG. Evaluation and Management of Penicillin Allergy: A Review. JAMA. 2019 Jan 15;321(2):188-199. doi: 10.1001/jama.2018.19283. PMID 30644987
- [Result] de Haan P, Bruynzeel DP, van Ketel WG. Onset of penicillin rashes: relation between type of penicillin administered and type of immune reactivity. Allergy. 1986 Jan;41(1):75-8. doi: 10.1111/j.1398-9995.1986.tb00279.x. PMID 2938516
- [Result] Blanca M, Romano A, Torres MJ, Fernandez J, Mayorga C, Rodriguez J, Demoly P, Bousquet PJ, Merk HF, Sanz ML, Ott H, Atanaskovic-Markovic M. Update on the evaluation of hypersensitivity reactions to betalactams. Allergy. 2009 Feb;64(2):183-93. doi: 10.1111/j.1398-9995.2008.01916.x. PMID 19133923
- [Result] Hjortlund J, Mortz CG, Skov PS, Bindslev-Jensen C. Diagnosis of penicillin allergy revisited: the value of case history, skin testing, specific IgE and prolonged challenge. Allergy. 2013 Aug;68(8):1057-64. doi: 10.1111/all.12195. Epub 2013 Jul 29. PMID 23889703
- [Result] Devillers L, Sicsic J, Delbarre A, Le Bel J, Ferrat E, Saint Lary O. General Practitioner trainers prescribe fewer antibiotics in primary care: Evidence from France. PLoS One. 2018 Jan 25;13(1):e0190522. doi: 10.1371/journal.pone.0190522. eCollection 2018. PMID 29370178